CLINICAL TRIAL: NCT05752617
Title: European Registry On Plaque ModifiCAtion in the STEMI Population (ROCA-STEMI)
Acronym: ROCA-STEMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Héctor Cubero Gallego, MD, PhD, Principal Investigator, Hospital del Mar
Other Study IDs: 2020/9525
Record Dates: First submitted 2023-02-15; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Calcified Coronary Lesions; ST Elevated Myocardial Infarction; Plaque Modification Technique
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an European prospective cohort study from February 2023 until February 2024. The investigators want to analyze the clinical success, efficacy and safety of consecutive patients who presented with ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI) for de novo heavily calcified culprit lesion using plaque modification devices before stent implantation.

DETAILED DESCRIPTION:
The ROCA-STEMI study is an European prospective cohort study from February 2023 until February 2024. The investigators want to analyze the clinical success, efficacy and safety of consecutive patients who presented with ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI) for de novo heavily calcified culprit lesion using plaque modification devices before stent implantation.

Clinical and angiographic endpoints will be defined according to the recommendations of the Academic Research Consortium. Academic Research Consortium represents a step toward standardization, facilitating the evaluation of the safety and effectiveness of devices.

Bleeding as a safety endpoint will be defined according to the Bleeding Academic Research Consortium. Major bleeding will be defined as Bleeding Academic Research Consortium types 3 and 5.

Severe coronary calcified lesion: Imaging evidence of severe calcium at the culprit lesion site was based on the angiographic presence of radio-opacities noted without cardiac motion before contrast injection involving both sides of the arterial wall in at least 1 location, or presence of ≥270° of calcium at 1 cross-section through IVUS.

Major adverse cardiovascular events (MACE): will be defined as the composite of cardiac death; MI; stroke, and revascularization, including percutaneous coronary intervention, and coronary artery bypass graft. Deaths will be regarded to be attributable to a cardiac cause unless a non-cardiac death could be confirmed.

Target lesion revascularization (TLR): will be defined as repeat PCI to treat the same lesion treated during the index procedure.

Target vessel revascularization (TVR): will be defined as PCI of a new severe lesion at another location other than the segment vessel treated at the index PCI.

Non-TVR: will be defined as PCI of a different vessel treated at the index procedure.

Target-lesion failure (TLF): will be defined as the composite of clinically-driven TLR, myocardial infarction, or cardiac death related to the target vessel.

Segment treated thrombosis (STT): is defined according to the Academic Research Consortium (ARC) definition as definite, probable, or possible and as early (0 to 30 days), late (31 to 360 days), or very late (>360 days).

Acute closure: is defined as the occurrence of new, severely reduced flow (grade 0 or 1, according to the Thrombolysis in Myocardial Infarction (TIMI) within the target vessel during the intervention that persists and requires another kind of treatment or results in MI or death.

Study device and procedures

Interventional procedure All coronary calcified lesions will be treated using at least one plaque-modification device. The concomitant use of other plaque-modification devices will be allowed in the presence of heavy calcium and at the operator's discretion.

Based on technology without balloon: rotational atherectomy (RA), orbital atherectomy (OA) and excimer laser coronary atherectomy (ELCA). Among devices based on technologies with balloon there are the cutting balloon, the scoring balloon, the coronary lithoplasty balloon (CL) and the super-high-pressure twin layer non-compliant (NC) balloon, OPN.

Cutting balloon and scoring balloon. The WOLVERINE cutting balloon (Boston Scientific, Marlborough, MA, United States) consists of a NC balloon with 3 micro-blades longitudinally arranged on its surface. Sequential inflation up to 6 atm is advisable. Other available devices are the AngioSculpt, Scoreflex, and NSE Alpha scoring balloons.

Shockwave Coronary IVL System. The lithoplasty balloon (LB) is a rapid-exchange balloon catheter with emitters that generate sonic waves to crack the calcium and to improve vessel compliance. The LB is inflated at calcified lesion level at a pressure of 4 atm and 1 Hz shockwaves are administered. Once the LB is on the lesion, it is connected to an external unit that generates pulsatile mechanical waves. The LB is initially inflated at a pressure of 4 atm and 10 pulses are administered (around 10 seconds are required). Then, the LB is inflated at a 6 atm pressure and then it is deflated to restore the flow. New cycles are then applied; a total of 8 therapies (80 pulses) per balloon and lesion can be administered. Due to its size, if the length of the lesion is > 12 mm, the LB can be repositioned to treat the lesion entirely.

Rotational atherectomy (RA): is an endovascular procedure to modify atherosclerotic plaque by advancing a diamond-coated rotating metal olive-shaped burr. The rotational speed recommended is between 135.000 rpm and 180.000 rpm. Decelerations > 5000 rpm should be avoided. The burr should be advanced gradually with easy back-and-forth moves and rotablation time should be < 20 seconds with pauses in between each cycle. Once rotablation has been performed, the olive-shaped burr is removed and the Dynaglide mode is activated.

Orbital atherectomy (OA): is an endovascular procedure to modify atherosclerotic plaque by using a diamond-coated crown whose mechanism of action consists of the antegrade and retrograde modification of the plaque.14-16 The OA mechanism of action is the elliptical rotation of the crown that gradually increases orbital diameter as rotation speed increases from 80.000 rpm to 120.000 rpm. The OA effect is time-dependent; 30 second-cycles are advisable with 30 second-pauses in between them. The continuous infusion of a lubricant solution (ViperSlide) is required to minimize thermal lesions during OA; also, 18 mL/min of fluid are administered to cool the device down and eliminate residue, thus reducing ischemia and distal embolization.

Excimer laser coronary atherectomy (ELCA): The Philips CVX-300 ELCA system uses xenon chloride and emits pulses of ultraviolet (UV) light at a 308-nm wavelength. The UV pulses generated only penetrate 50 μm deep, which disintegrates the calcified plaque through a mechanism of ablation without damage to the middle or adventitia layers.29,30 There are 4 different sizes of ELCA monorail catheter available (0.9, 0.14, 1.7 and 2.0 mm) that can be advanced on a 0.014 in guidewire. The right size is selected on a 0.5:0.6 ratio between catheter and vessel. Slowly moving the device forward promotes an increased luminal gain at lesion level. The number of pulses, length and total time of ELCA treatment should be individualized depending on the characteristics of the lesion. The particles generated have a diameter < 10 μm so they are reabsorbed by the reticuloendothelial system, thus avoiding microvascular obstruction.

The implantation of a drug-eluting stent (DES) is then performed at the discretion of the operator along with high-pressure (>16 atm) postdilation. Dual-antiplatelet therapy will be administered following the established clinical practice guidelines.

Clinical and angiographic data Clinical data and clinical events will be investigator-reported through an electronic case report form (eCRF). Detailed outcome definitions have been described previously.

Angiographic analysis the presence of severe coronary calcification was evaluated, based on coronary angiography, during the index procedure by each investigator at the participating centers.

Ethics Aspects The study will be conducted according to the ethical principles derived from the Declaration of Helsinki (Fortaleza, Brazil, October 2013), ISO 14155, and clinical practice guidelines. In addition, the study will be conducted according to the protocol of Good Clinical Practice (GCP) following the International Conference on Harmonization (ICH) guidelines and regulatory requirements for participating institutions. The study protocol was approved by the Institutional Ethics Committee and the hospital's research commission. Once a patient has been identified as a candidate for participation in the study (meeting all inclusion criteria and none exclusion criteria), and after duly informing the patient about the characteristics of the study, an informed consent will be signed and recorded in the corresponding file of the center's investigator. Baseline demographics, procedural features, clinical outcomes and follow-up data will be collected by the coinvestigators at each institution through dedicated electronic case report form (e-CRF).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with a STEMI
* Primary percutaneous coronary intervention
* De-novo culprit lesion in a native coronary artery
* Severe calcification of the target lesion or its equivalent (balloon uncrossable or undilatable lesion) (See Definitions 4.4)
* Mandatory use of a plaque modification device to treat the culprit lesion (See Study device and procedures 4.5)
* The patient or legal representative signing an informed written consent

Exclusion Criteria:

* The target vessel had a stent from a previous PCI
* The target lesion was treated as a staged procedure
* Pregnant women
* Terminally ill patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The ROCA-STEMI study is an European prospective cohort study from February 2023 until February 2024. We want to analyze the clinical success, efficacy and safety of consecutive patients who presented with ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI) for de novo heavily calcified culprit lesion using plaque modification devices before stent implantation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure | 12 months
  The occurrence of cardiac death, target vessel myocardial infraction and target vessel revascularization.

SECONDARY OUTCOMES:
Cardiac death | 12 months
  Death that could not be attributed to a noncardiac etiology was considered cardiac death.
Major Adverse Cardiac Events (MACE) | 12 months
  Major Adverse Cardiac Events (MACE) at 12 months (death, re-infarction, acute cardiovascular disease, hemorrhagy and/or stent thrombosis).
Target vessel revascularization | 12 months
  Target vessel revascularization was defined as repeated revascularization by PCI or surgery of the target vessel.
Target lesion revascularization | 12 months
  Target lesion revascularization was defined as any revascularization procedure performed at the site of the treated lesion associated with clinical and/or objective evidence of inducible myocardial ischemia.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

REFERENCES:
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO. 2018 ESC/EACTS Guidelines on myocardial revascularization. EuroIntervention. 2019 Feb 20;14(14):1435-1534. doi: 10.4244/EIJY19M01_01. No abstract available. PMID 30667361
- [Background] Otsuka F, Sakakura K, Yahagi K, Joner M, Virmani R. Has our understanding of calcification in human coronary atherosclerosis progressed? Arterioscler Thromb Vasc Biol. 2014 Apr;34(4):724-36. doi: 10.1161/ATVBAHA.113.302642. Epub 2014 Feb 20. PMID 24558104
- [Background] Bourantas CV, Zhang YJ, Garg S, Iqbal J, Valgimigli M, Windecker S, Mohr FW, Silber S, Vries Td, Onuma Y, Garcia-Garcia HM, Morel MA, Serruys PW. Prognostic implications of coronary calcification in patients with obstructive coronary artery disease treated by percutaneous coronary intervention: a patient-level pooled analysis of 7 contemporary stent trials. Heart. 2014 Aug;100(15):1158-64. doi: 10.1136/heartjnl-2013-305180. Epub 2014 May 20. PMID 24846971
- [Background] Witzenbichler B, Maehara A, Weisz G, Neumann FJ, Rinaldi MJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Brodie BR, Stuckey TD, Mazzaferri EL Jr, Xu K, Parise H, Mehran R, Mintz GS, Stone GW. Relationship between intravascular ultrasound guidance and clinical outcomes after drug-eluting stents: the assessment of dual antiplatelet therapy with drug-eluting stents (ADAPT-DES) study. Circulation. 2014 Jan 28;129(4):463-70. doi: 10.1161/CIRCULATIONAHA.113.003942. Epub 2013 Nov 26. PMID 24281330
- [Background] Barbato E, Shlofmitz E, Milkas A, Shlofmitz R, Azzalini L, Colombo A. State of the art: evolving concepts in the treatment of heavily calcified and undilatable coronary stenoses - from debulking to plaque modification, a 40-year-long journey. EuroIntervention. 2017 Aug 25;13(6):696-705. doi: 10.4244/EIJ-D-17-00473. PMID 28844031
- [Background] De Maria GL, Scarsini R, Banning AP. Management of Calcific Coronary Artery Lesions: Is it Time to Change Our Interventional Therapeutic Approach? JACC Cardiovasc Interv. 2019 Aug 12;12(15):1465-1478. doi: 10.1016/j.jcin.2019.03.038. PMID 31395217
- [Background] Shavadia JS, Vo MN, Bainey KR. Challenges With Severe Coronary Artery Calcification in Percutaneous Coronary Intervention: A Narrative Review of Therapeutic Options. Can J Cardiol. 2018 Dec;34(12):1564-1572. doi: 10.1016/j.cjca.2018.07.482. Epub 2018 Aug 14. PMID 30527144
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Abdel-Wahab M, Richardt G, Joachim Buttner H, Toelg R, Geist V, Meinertz T, Schofer J, King L, Neumann FJ, Khattab AA. High-speed rotational atherectomy before paclitaxel-eluting stent implantation in complex calcified coronary lesions: the randomized ROTAXUS (Rotational Atherectomy Prior to Taxus Stent Treatment for Complex Native Coronary Artery Disease) trial. JACC Cardiovasc Interv. 2013 Jan;6(1):10-9. doi: 10.1016/j.jcin.2012.07.017. Epub 2012 Dec 19. PMID 23266232
- [Background] Abdel-Wahab M, Toelg R, Byrne RA, Geist V, El-Mawardy M, Allali A, Rheude T, Robinson DR, Abdelghani M, Sulimov DS, Kastrati A, Richardt G. High-Speed Rotational Atherectomy Versus Modified Balloons Prior to Drug-Eluting Stent Implantation in Severely Calcified Coronary Lesions. Circ Cardiovasc Interv. 2018 Oct;11(10):e007415. doi: 10.1161/CIRCINTERVENTIONS.118.007415. PMID 30354632
- [Background] Kawamoto H, Latib A, Ruparelia N, Ielasi A, D'Ascenzo F, Pennacchi M, Sardella G, Garbo R, Meliga E, Moretti C, Rossi ML, Presbitero P, Magri CJ, Nakamura S, Colombo A, Boccuzzi GG. In-hospital and midterm clinical outcomes of rotational atherectomy followed by stent implantation: the ROTATE multicentre registry. EuroIntervention. 2016 Dec 20;12(12):1448-1456. doi: 10.4244/EIJ-D-16-00386. PMID 27998836
- [Background] Parikh K, Chandra P, Choksi N, Khanna P, Chambers J. Safety and feasibility of orbital atherectomy for the treatment of calcified coronary lesions: the ORBIT I trial. Catheter Cardiovasc Interv. 2013 Jun 1;81(7):1134-9. doi: 10.1002/ccd.24700. Epub 2013 Mar 5. PMID 23460596
- [Background] Chambers JW, Feldman RL, Himmelstein SI, Bhatheja R, Villa AE, Strickman NE, Shlofmitz RA, Dulas DD, Arab D, Khanna PK, Lee AC, Ghali MG, Shah RR, Davis TP, Kim CY, Tai Z, Patel KC, Puma JA, Makam P, Bertolet BD, Nseir GY. Pivotal trial to evaluate the safety and efficacy of the orbital atherectomy system in treating de novo, severely calcified coronary lesions (ORBIT II). JACC Cardiovasc Interv. 2014 May;7(5):510-8. doi: 10.1016/j.jcin.2014.01.158. PMID 24852804
- [Background] Lee M, Genereux P, Shlofmitz R, Phillipson D, Anose BM, Martinsen BJ, Himmelstein SI, Chambers JW. Orbital atherectomy for treating de novo, severely calcified coronary lesions: 3-year results of the pivotal ORBIT II trial. Cardiovasc Revasc Med. 2017 Jun;18(4):261-264. doi: 10.1016/j.carrev.2017.01.011. Epub 2017 Jan 23. PMID 28162989
- [Background] Ali ZA, Brinton TJ, Hill JM, Maehara A, Matsumura M, Karimi Galougahi K, Illindala U, Gotberg M, Whitbourn R, Van Mieghem N, Meredith IT, Di Mario C, Fajadet J. Optical Coherence Tomography Characterization of Coronary Lithoplasty for Treatment of Calcified Lesions: First Description. JACC Cardiovasc Imaging. 2017 Aug;10(8):897-906. doi: 10.1016/j.jcmg.2017.05.012. PMID 28797412
- [Background] Brinton TJ, Ali ZA, Hill JM, Meredith IT, Maehara A, Illindala U, Lansky A, Gotberg M, Van Mieghem NM, Whitbourn R, Fajadet J, Di Mario C. Feasibility of Shockwave Coronary Intravascular Lithotripsy for the Treatment of Calcified Coronary Stenoses. Circulation. 2019 Feb 5;139(6):834-836. doi: 10.1161/CIRCULATIONAHA.118.036531. No abstract available. PMID 30715944
- [Background] Ali ZA, Nef H, Escaned J, Werner N, Banning AP, Hill JM, De Bruyne B, Montorfano M, Lefevre T, Stone GW, Crowley A, Matsumura M, Maehara A, Lansky AJ, Fajadet J, Di Mario C. Safety and Effectiveness of Coronary Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Stenoses: The Disrupt CAD II Study. Circ Cardiovasc Interv. 2019 Oct;12(10):e008434. doi: 10.1161/CIRCINTERVENTIONS.119.008434. Epub 2019 Sep 25. PMID 31553205
- [Background] Wang X, Matsumura M, Mintz GS, Lee T, Zhang W, Cao Y, Fujino A, Lin Y, Usui E, Kanaji Y, Murai T, Yonetsu T, Kakuta T, Maehara A. In Vivo Calcium Detection by Comparing Optical Coherence Tomography, Intravascular Ultrasound, and Angiography. JACC Cardiovasc Imaging. 2017 Aug;10(8):869-879. doi: 10.1016/j.jcmg.2017.05.014. PMID 28797408
- [Background] Hill JM, Kereiakes DJ, Shlofmitz RA, Klein AJ, Riley RF, Price MJ, Herrmann HC, Bachinsky W, Waksman R, Stone GW; Disrupt CAD III Investigators. Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Artery Disease. J Am Coll Cardiol. 2020 Dec 1;76(22):2635-2646. doi: 10.1016/j.jacc.2020.09.603. Epub 2020 Oct 15. PMID 33069849
- [Background] Stolker JM, Cohen DJ, Kennedy KF, Pencina MJ, Lindsey JB, Mauri L, Cutlip DE, Kleiman NS; Evaluation of Drug-Eluting Stents and Ischemic Events (EVENT) Investigators. Repeat revascularization after contemporary percutaneous coronary intervention: an evaluation of staged, target lesion, and other unplanned revascularization procedures during the first year. Circ Cardiovasc Interv. 2012 Dec;5(6):772-82. doi: 10.1161/CIRCINTERVENTIONS.111.967802. Epub 2012 Oct 23. PMID 23093553
- [Background] Mauri L, Bonan R, Weiner BH, Legrand V, Bassand JP, Popma JJ, Niemyski P, Prpic R, Ho KK, Chauhan MS, Cutlip DE, Bertrand OF, Kuntz RE. Cutting balloon angioplasty for the prevention of restenosis: results of the Cutting Balloon Global Randomized Trial. Am J Cardiol. 2002 Nov 15;90(10):1079-83. doi: 10.1016/s0002-9149(02)02773-x. PMID 12423707
- [Background] Cubero-Gallego H, Gonzalo N, Tizon-Marcos H, Salvatella N, Garcia-Guimaraes M, Negrete A, McInerney A, Millan R, Vaquerizo B. Primary Angioplasty of Calcified Coronary Lesions Using Coronary Lithotripsy in Acute ST-Segment Elevation Myocardial Infarction. J Invasive Cardiol. 2021 Dec;33(12):E970-E973. doi: 10.25270/jic/21.00015. Epub 2021 Nov 11. PMID 34783676
- [Background] Sharma SK, Tomey MI, Teirstein PS, Kini AS, Reitman AB, Lee AC, Genereux P, Chambers JW, Grines CL, Himmelstein SI, Thompson CA, Meredith IT, Bhave A, Moses JW. North American Expert Review of Rotational Atherectomy. Circ Cardiovasc Interv. 2019 May;12(5):e007448. doi: 10.1161/CIRCINTERVENTIONS.118.007448. PMID 31084239
- [Background] Barbato E, Carrie D, Dardas P, Fajadet J, Gaul G, Haude M, Khashaba A, Koch K, Meyer-Gessner M, Palazuelos J, Reczuch K, Ribichini FL, Sharma S, Sipotz J, Sjogren I, Suetsch G, Szabo G, Valdes-Chavarri M, Vaquerizo B, Wijns W, Windecker S, de Belder A, Valgimigli M, Byrne RA, Colombo A, Di Mario C, Latib A, Hamm C; European Association of Percutaneous Cardiovascular Interventions. European expert consensus on rotational atherectomy. EuroIntervention. 2015 May;11(1):30-6. doi: 10.4244/EIJV11I1A6. PMID 25982648
- [Background] Ho PC. Rotational coronary atherectomy in acute ST-segment elevation myocardial infarction. J Interv Cardiol. 2005 Aug;18(4):315-8. doi: 10.1111/j.1540-8183.2005.00057.x. PMID 16115167
- [Background] Mokabberi R, Blankenship JC. Rotational atherectomy to facilitate stent expansion after deployment in ST-segment-elevation myocardial infarction. Am Heart Hosp J. 2010 Summer;8(1):66-9. doi: 10.15420/ahhj.2010.8.1.66. PMID 21194056
- [Background] Appelman YE, Piek JJ, Strikwerda S, Tijssen JG, de Feyter PJ, David GK, Serruys PW, Margolis JR, Koelemay MJ, Montauban van Swijndregt EW, Koolen JJ. Randomised trial of excimer laser angioplasty versus balloon angioplasty for treatment of obstructive coronary artery disease. Lancet. 1996 Jan 13;347(8994):79-84. doi: 10.1016/s0140-6736(96)90209-3. PMID 8538345
- [Background] Stone GW, de Marchena E, Dageforde D, Foschi A, Muhlestein JB, McIvor M, Rizik D, Vanderlaan R, McDonnell J. Prospective, randomized, multicenter comparison of laser-facilitated balloon angioplasty versus stand-alone balloon angioplasty in patients with obstructive coronary artery disease. The Laser Angioplasty Versus Angioplasty (LAVA) Trial Investigators. J Am Coll Cardiol. 1997 Dec;30(7):1714-21. doi: 10.1016/s0735-1097(97)00387-2. PMID 9385898